CLINICAL TRIAL: NCT02324777
Title: A Randomized Double Blind Placebo Controlled, Proof-of-concept, Crossover Clinical Trial of Vapourized Cannabis in Adults With Painful Osteoarthritis of the Knee
Brief Title: Cannabinoid Profile Investigation of Vapourized Cannabis in Patients With Osteoarthritis of the Knee
Acronym: CAPRI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prairie Plant Systems Inc. (Industry)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Dalhousie University (Other); Algorithme Pharma Inc (Industry); Research Institute of the McGill University Health Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PPS001
Record Dates: First submitted 2014-12-05; First posted 2014-12-24 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- CanniMed™ DPF-I Volcano® Vapourization (Experimental): Using the Volcano® Medic, a dose of 100 mg of finely ground herbal cannabis drug product formulation (DPF) with a potency specification similar to CanniMed™ 22·1 product, of 21.9% w/w total THC and 0.8% w/w total CBD is vapourized and inhaled by study subjects.
  Interventions: Drug: Cannabis; Device: Volcano® Medic Vapourizer
- CanniMed™ DPF-II Volcano® Vapourization (Experimental): Using the Volcano® Medic, a dose of 100 mg of finely ground herbal cannabis drug product formulation with a potency specification the same as the CanniMed™ 15·5 product, of 15.0% w/w total THC and 5.0% w/w total CBD is vapourized and inhaled by study subjects.
  Interventions: Drug: Cannabis; Device: Volcano® Medic Vapourizer
- CanniMed™ DPF-III Volcano® Vapourization (Experimental): Using the Volcano® Medic, a dose of 100 mg of finely ground herbal cannabis drug product formulation with a potency specification the same as CanniMed™ 9·9 product, of 9.0% w/w total THC and 9.5% w/w total CBD is vapourized and inhaled by study subjects.
  Interventions: Drug: Cannabis; Device: Volcano® Medic Vapourizer
- CanniMed™ DPF-IV Volcano® Vapourization (Experimental): Using the Volcano® Medic, a dose of 100 mg of finely ground herbal cannabis drug product formulation with a potency specification similar to CanniMed™ 4·10 product, of 3.8% w/w total THC and 10.0% w/w total CBD is vapourized and inhaled by study subjects.
  Interventions: Drug: Cannabis; Device: Volcano® Medic Vapourizer
- CanniMed™ DPF-V Volcano® Vapourization (Experimental): Using the Volcano® Medic, a dose of 100 mg of finely ground herbal cannabis drug product formulation with a potency specification similar to CanniMed™ 1·13 product profile of 0.6% w/w total THC and 13.0% w/w total CBD is vapourized and inhaled by study subjects.
  Interventions: Drug: Cannabis; Device: Volcano® Medic Vapourizer
- CanniMed™ DPF-P Volcano® Vapourization (Placebo Comparator): Using the Volcano® Medic, a dose of 100 mg of ethanol extracted DPF-V, reducing the potency profile to <0.3% w/w total THC and <0.3% w/w total CBD (comparable to the threshold levels described for "industrial hemp", as per the Canadian Industrial Hemp Regulations (SOR/98-156), is vapourized and inhaled by study subjects.
  Interventions: Drug: Cannabis; Device: Volcano® Medic Vapourizer

INTERVENTIONS:
Drug: Cannabis — Cannabis sativa L. subsp. indica, variety indica blends of flowering heads that have been air-dried, milled, destemmed and fine ground, stored in glass vials with aluminum caps in 100 mg dose size.
  Other Names: Marijuana; Marihuana; CanniMed™
Device: Volcano® Medic Vapourizer — Volcano® Medic vapourizer is licensed for medical administration of cannabis in Canada March 2010 (Licence No. 82405).
  The contents of a vial of drug product formulation will be transferred to the Volcano® Medic's filling chamber (sample-holder) equipped top and bottom with fine wire mesh to retain the finely ground material. The filling chamber will be placed atop the main body of the unit and then have a, 12.5 L, heat-resistant Medic Valve balloon affixed. Active components are vapourized at 190 °C. The ensuing vapour is captured in the balloon and inhaled by the study subject using a standardized inhalation technique.

SUMMARY:
Primary Objective:

- To determine the analgesic dose-response characteristics of vapourized cannabinoids with varying degrees of delta-9-tetrahydrocannabiol (THC)/ Cannabidiol (CBD) ratios.

Secondary Objectives:

* To compare functional changes and patient preferences of different cannabinoid (THC, CBD) profiles in patients with OA (Osteoarthritis);
* To describe the Pharmacokinetics (PK) of vapourized cannabis of differing cannabinoid profiles in patients with OA;
* To explore the short term safety of vapourized cannabis with different cannabinoid profiles.
* To describe the incidence and severity of psychoactive events.

DETAILED DESCRIPTION:
A Phase IIa randomized double blind placebo controlled crossover trial (RCT) using six different herbal cannabis drug product formulations prepared by the Sponsor, Prairie Plant Systems Inc. An initial screening period (minimum one week) will be completed for pain assessment and determination of eligibility. After screening, eligible subjects will be randomly assigned to receive all 6 different formulations in a random order.

The study will be conducted using six periods of 7 days duration, with each period consisting of one day of exposure and 6 days of washout from study drug. The study will therefore take 6 weeks to be completed for each enrolled subject with an additional week for adverse event monitoring after the final study exposure. Total time in study may therefore be a maximum of nine weeks (including screening).

Adult subjects (age ≥50y) will be recruited with chronic (>3 months) moderate to severe pain (pain score ≥40/100 on visual analogue scale) due to primary osteoarthritis (OA) of the knee as defined by American College of Rheumatology (ACR) criteria. Target enrolment for this study is 36 (18 from each site).

The study will be conducted at the Alan Edwards Pain Management Unit of the McGill University Health Centre, in Montreal, Quebec, Canada and the Pain Management Unit at the Queen Elizabeth II Health Sciences Centre in Halifax, Nova Scotia, Canada. A dedicated ventilated room is available at these sites for cannabinoid inhalation studies as used in prior evaluation trials on medicinal cannabis.

All subjects meeting eligibility criteria after the screening period will be randomized to receive all 6 herbal cannabis drug product formulations in a randomly assigned order of treatment between Clinical Visit (CV) 2 and CV7.

A washout period of 6 days is proposed between the six different treatment periods. This will allow the pharmacological effects of each dose to be minimized prior to each subsequent dosing period to avoid confounding.

Throughout the study all subjects will remain on their stable (pharmacological and non-pharmacological) treatment regimen.

Throughout the study, subjects will be blinded to the treatment they are receiving. Once a subject has been randomized, the investigator and the subject, as well as all staff involved in the conduct or management of the study will be blinded to the treatment assignment. All dosing will be via the Volcano® Medic vapourizer (licensed for medical administration of cannabis in Canada March 2010; Licence No. 82405) and both the nurse and the patient will be familiarized with its instruction manual.

The study nurse will prepare the dose for the subject. After opening the vial of drug product formulation, its contents will be transferred to the Volcano® Medic's filling chamber (sample-holder) equipped top and bottom with fine wire mesh to retain the finely ground material. The filling chamber will be placed atop the main body of the unit and then have a, 12.5 L, heat-resistant Medic Valve balloon affixed to it (this balloon will be housed within an opaque bag that is required to ensure blinding because the placebo generates little in the way of visible vapour). Active components (THCA and CBDA decarboxylated to THC and CBD) will be vapourized out of the herbal material by a stream of hot air with an exact, predefined temperature (190 °C). The ensuing vapour will be captured in the balloon. After filling has been completed (35 seconds), a mouthpiece will be attached to the balloon for inhalation of the vapour by the study subject. The total contents of the balloon will be inhaled over five minutes by using a standardized inhalation technique. Immediately after the bag has been removed from the Volcano® Medic, inhalation will be according to the following regimen:

1. Inhale for 4 seconds
2. Hold breath for 6 seconds
3. Exhale and breathe normally for 20 seconds
4. Repeat this inhale-hold-breathe cycle (30 seconds) until the bag has been evacuated.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic (primary) OA of the knee as defined by American College of Rheumatology criteria
2. Age ≥50 years
3. Numerical Rating Scale (NRS) Pain intensity score ≥ 4 (on a 0-10 scale)
4. Stable medication and treatment regimen
5. Open to Canadian Residents only

Exclusion Criteria:

1. Pregnant/nursing
2. BMI >39kg/m2
3. Secondary causes of OA
4. Stage IV OA of the knee
5. Significant other cause of pain (e.g. fibromyalgia, CRPS)
6. Significant cardiac, neurological, psychiatric or respiratory disease
7. Joint infiltration in 30 days prior to trial or during study
8. Positive urine screen for THC

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Total pain reduction of vapourized cannabinoids with varying degrees of THC/CBD ratios in patients with painful OA of the knee. | 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes post-dose
  The main efficacy endpoint is pain reduction, calculated as a change in pain intensity (VAS pain intensity) following each exposure. A Total Pain Reduction (TOTPAR) score is calculated from repeated VAS pain scores taken immediately before (baseline) and every 15 minutes after exposure for the first hour then half-hourly for the remaining two hours after treatment exposure (treatment). The treatment VAS pain intensity scores are then subtracted from the baseline VAS pain intensity to generate a pain relief score for each time point. The sum of pain relief scores from each time point is used to generate a 3-hour Total Pain Reduction (TOTPAR-3) score for each exposure.

SECONDARY OUTCOMES:
Pain, stiffness, physical, social and emotional functional outcomes of vapourized cannabis with varying degrees of THC/CBD ratios in patients with painful OA of the knee. | Up to 6 weeks
  Pain and functional outcomes will be measured using the Western Ontario and McMaster Osteoarthritis Index (WOMAC).
  The WOMAC Osteoarthritis Index is a 24-item instrument that assesses the three dimensions of pain, disability and joint stiffness in studies of knee and hip osteoarthritis. The WOMAC Osteoarthritis Index will be completed by the subject at Visit 2-8.
Pharmacokinetics profile of 7 plasma cannabinoid metabolites from vapourized cannabis of differing cannabinoid profiles in patients with OA. | 0, 15, 30, 60, 120 and 180 minutes post-dose
  Pharmacokinetic analysis encompasses an assay validated for: Δ9-tetrahydrocannabinol (THC); 11-nor-Δ9-tetrahydrocannabinol-9-carboxylic acid (11-nor-Δ9-THC-9-COOH); 11-hydroxy-Δ9-tetrahydrocannabinol (11-OH-THC); cannabinol (CBN); cannabidiol (CBD); and qualified for: Δ9-tetrahydrocannabinolic acid (THCA); cannabidiolic acid (CBDA).
  Blood will be taken prior to inhalation (T = 0) and at 2, 30, 60, and 180 minutes after each exposure for pharmacokinetic assessments of plasma cannabinoid levels. These intervals have been used to evaluate PK of vapourized cannabis in healthy volunteers (Abrams, et al., 2007).
Changes in blood pressure from baseline | Up to 7 weeks
  Resting/sitting and postural change in blood pressure are assessed at screening and at each subsequent clinical visit where the interventions are used to gauge changes and acute or sustained changes during the course of treatment. Sitting and postural change in BP are taken at 0, 30, 60, 90, 120, 150, and 180 minutes post-dose.
Changes in heart rate (HR) from baseline | Up to 7 weeks
  Sitting heart rates are assessed at screening and at each subsequent clinical visit where the interventions are used to gauge changes and acute or sustained changes during the course of treatment. Sitting HR is taken at 0, 30, 60, 90, 120, 150, and 180 minutes post-dose.
Blood chemistry - liver function | Up to 7 weeks
  Blood is taken at screening, and then for each clinical visit where the interventions are used at T = 0 (prior to inhalation) and at T = 180 minutes (end of study visit) for aspartate aminotransferase (AST) or serum glutamic oxaloacetic transaminase (SGOT). Inclusion criteria for candidates is AST < 3X normal (normal = 5 - 40 units per litre of serum). Change from baseline at screening and per visit with intervention will be assessed for short term liver changes following a single exposure to differing levels of inhaled THC and/or CBD.
Blood chemistry - renal function | Up to 7 weeks
  Blood is taken at screening, and then for each clinical visit where the interventions are used at T = 0 (prior to inhalation) and at T = 180 minutes (end of study visit) for serum creatinine. Inclusion criteria for candidates is serum creatinine < 133 μmol/. Change from baseline at screening and per visit with intervention will be assessed for short term renal changes following a single exposure to differing levels of inhaled THC and/or CBD.
Hematology - hematocrit level (complete blood count) | Up to 7 weeks
  Blood is taken at screening, and then for each clinical visit where the interventions are used at T = 0 (prior to inhalation) and at T = 180 minutes (end of study visit) for hematocrit level (or CBC). Inclusion criteria for candidates is CBC > 35%. Change from baseline at screening and per visit with intervention will be assessed for short term hematological changes following a single exposure to differing levels of inhaled THC and/or CBD.
Cannabinoid urine analysis at screening and for washout confirmation | Up to 7 weeks
  Urine analysis (THC = 50 mg/mL) will be performed at each clinical visit to gauge cannabinoid clearance prior to the interventions and to ensure that washout between interventions is maintained as each dose should not produce a sustained 1 week urine result.
Psychoactive adverse events | Up to 6 weeks
  A Psychoactive Adverse Event checklist will be administered by the Research Nurse to the participant to report on any changes in their emotional state (such as anxiety, panic, paranoia, depersonalization, mood alteration and altered perceptions etc) every 15 minutes after exposure for the first hour then half-hourly for the remaining two hours.
Patient global rating of preference for each cannabis preparation. | Up to 6 weeks
  Patient global rating of preference for each cannabis preparation will be measured using a VAS (drug liking 0: Do not like at all; 100: really like a lot) after each exposure, and a global ranking after all six exposures have been completed.
Visual Analog Scale (VAS) feelings of drug effect | Up to 6 weeks
  The VAS for feelings of drug effect is a horizontal line measurement of 100mm with Anchors of 0 = not high at all and 100 = most high ever. Subjects mark their Feeling of Drug Effect by placing a vertical line through the horizontal line to indicate how "high" they are feeling NOW.
  The VAS for Feelings of Drug Effect will be completed by the subject at each intervention visit; taken at 15 minute intervals after exposure for the first hour then half-hourly for the remaining two hours.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ware, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Mary Lynch, MD, Principal Investigator — Queen Elizabeth II Health Science Centre
Locations (2):
- Canada (2):
  - Pain Management Unit, Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Montreal General Hospital - McGill University Health Centre, Montreal, Quebec

REFERENCES:
- [Background] Abrams DI, Vizoso HP, Shade SB, Jay C, Kelly ME, Benowitz NL. Vaporization as a smokeless cannabis delivery system: a pilot study. Clin Pharmacol Ther. 2007 Nov;82(5):572-8. doi: 10.1038/sj.clpt.6100200. Epub 2007 Apr 11. PMID 17429350
- See also: WOMAC Osteoarthritis Index — http://www.womac.org/contact/index.htm
- See also: CanniMed Ltd. - Canadian Licensed Medical Marijuana Supplier — http://www.cannimed.ca